CLINICAL TRIAL: NCT03112213
Title: CONIFER (Characterization of NSAID Intake for Established Rheumatoid Arthritis)
Brief Title: Characterization of Non-Steroidal Anti-Inflammatory Drug (NSAID) Intake in Rheumatoid Arthritis (RA) Participants on Tocilizumab (RoACTEMRA®) Treatment
Acronym: CONIFER
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML30088
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants With RA: Participants with RA who are being treated with tocilizumab and NSAIDs will be observed for approximately 6 months to evaluate the quantitative pattern of NSAID use and the impact of treatment with tocilizumab on NSAID use.
  Interventions: Drug: Tocilizumab; Drug: NSAIDs

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab (SC or IV) will be prescribed according to local clinical practice and the SPC.
  Other Names: RoACTEMRA®
Drug: NSAIDs — Participants may receive NSAIDs, as prescribed by the treating physician or by self medication. Study protocol does not enforce any particular NSAID.

SUMMARY:
This nationwide, multicenter, single arm, prospective, non-interventional study will evaluate the quantitative pattern of NSAID use and the impact of treatment with tocilizumab on NSAID use in a representative cohort of participant with moderate to severe active RA who have either responded inadequately to, or who were intolerant to previous therapy with one or more synthetic disease modifying anti-rheumatic drug (sDMARD), and for whom the physician has made the individual decision to initiate tocilizumab (subcutaneous [SC] or intravenous [IV]) as first biological disease modifying anti-rheumatic drug (DMARD) therapy according to the summary of product characteristics (SPC).

ELIGIBILITY:
Inclusion Criteria:

* Participants with moderate to severe active RA who have either responded inadequately to, or who were intolerant to, previous therapy with one or more sDMARDs and for whom the physician has made the individual decision to be treated with tocilizumab (SC or IV)
* Current users of NSAIDs due to RA as assessed by the physician

Exclusion Criteria:

* Contraindications to treatment with tocilizumab as per SPC
* Prior therapy with tocilizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2017-01-12 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2018-07-17 (Actual)

PRIMARY OUTCOMES:
Amount of NSAIDs Used During 14 Days Prior to First Tocilizumab Administration | Day -14 to Day 0 (Baseline)
Amount of NSAIDs Used During 14 Days After 6-8 Weeks of Tocilizumab Administration | 14 days after 6-8 weeks of tocilizumab administration
Amount of NSAIDs Used During 14 Days After 12-16 Weeks of Tocilizumab Administration | 14 days after 12-16 weeks of tocilizumab administration
Percentage of Participants by NSAIDs Dose Categories (Low-Dose and High-Dose) During 14 Days Prior to First Tocilizumab Administration | Day -14 to Day 0 (Baseline)
  NSAIDs high-dose refers to mean defined daily dose (DDD) greater than (>) 100 percent (%) and low-dose refers to mean DDD lesser than or equal to (</=) 100%.
Percentage of Participants by NSAIDs Dose Categories (Low-Dose and High-Dose) During 14 Days After 6-8 Weeks of Tocilizumab Administration | 14 days after 6-8 weeks of tocilizumab administration
  NSAIDs high-dose refers to mean DDD >100% and low-dose refers to mean DDD </=100%.
Percentage of Participants by NSAIDs Dose Categories (Low-Dose and High-Dose) During 14 Days After 12-16 Weeks of Tocilizumab Administration | 14 days after 12-16 weeks of tocilizumab administration
  NSAIDs high-dose refers to mean DDD >100% and low-dose refers to mean DDD </=100%.

SECONDARY OUTCOMES:
Percentage of Participants Who Take NSAIDs | Day -14 up to approximately Day 126
Average Daily Dose of NSAIDs | Day -14 up to approximately Day 126
Percentage of Participants Who Take NSAIDs Despite the Presence of Contraindications and Risk Factors | Day -14 up to approximately Day 126
Percentage of Participants Who do not Take Gastro-Protection (Proton-Pump Inhibitors [PPIs]) While Using NSAIDs | Day -14 up to approximately Day 126
Percentage of NSAID-Prescribers | Day -14 up to approximately Day 126
Percentage of NSAID Self-Medication | Day -14 up to approximately Day 126
Percentage of Participants Using NSAIDs by Disease Activity | Day -14 up to approximately Day 126
Percentage of Participants Using NSAIDs by Disease Duration | Day -14 up to approximately Day 126
Percentage of Participants Using NSAIDs by Health Assessment Questionnaire-Disability Index (HAQ-DI) Score | Day -14 up to approximately Day 126
HAQ-DI Score | Screening (up to 28 days prior to first tocilizumab administration); Day 0 (Baseline); Weeks 6-8; Weeks 12-16
Disease Activity Score Based on 28 Joints (DAS28) | Screening (up to 28 days prior to first tocilizumab administration); Day 0 (Baseline); Weeks 6-8; Weeks 12-16
Clinical Disease Activity Index (CDAI) Score | Screening (up to 28 days prior to first tocilizumab administration); Day 0 (Baseline); Weeks 6-8; Weeks 12-16
Simplified Disease Activity Index (SDAI) Score | Screening (up to 28 days prior to first tocilizumab administration); Day 0 (Baseline); Weeks 6-8; Weeks 12-16
Percentage of Participants With Adverse Events (AEs) | From Baseline up to approximately Week 28

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (27):
- Germany (27):
  - Rheumazentrum Kupka, Altenburg
  - Praxis für Rheumatologie., Amberg
  - Kerckhoff-Klinik; Rheumatologie&klin.Immunologie, Bad Nauheim
  - Charité Campus Mitte, Med.Klinik, Rheumatologie und Klinische Immunologie, Berlin
  - Praxis für Innere Medizin - Rheumatologie, Berlin
  - Rheuma Praxis Berlin Sven Remstedt, Berlin
  - Praxis Dr. Silke Zinke, Berlin
  - Schwerpunktpraxis für Rheumatologie und klinische Immunologie an den Kreiskliniken, Burghausen
  - Universitätsklinikum "Carl Gustav Carus"; Medizinische Klinik III, Dresden
  - Praxis Dr. med. Semmler; Facharzt für Innere Medizin, Güstrow
  - Dres.Karin Babinsky und Anke Liebhaber, Halle
  - Rheumatologische Schwerpunktpraxis, Hanover
  - Rheumapraxis PD Dr.med. Bernhard Heilig, Heidelberg
  - Rheumatologische Facharztpraxis Maren Sieburg, Magdeburg
  - Praxis für Innere Medizin und Rheumatologie, Mansfeld
  - Praxis Prof. Dr.med. Herbert Kellner, München
  - Praxiszentrum St. Bonifatius, München
  - Rheumatologische Praxis, Neubrandenburg
  - Rheumazentrum Neuss Dres. Irmgard Gürtler und Christoph Volberg, Neuss
  - Praxis Dr.med. Christoph Volberg, Neuss
  - Praxis Dr. Albert, Offenburg
  - Praxis für Rheumatologie Dr. med. Hauke E. Heintz, Poppenbüttel
  - Knappschaftsklinikum Saar GmbH, Krankenhaus Püttlingen, Püttlingen
  - Rheumazentrum Ratingen - Studienambulanz, Ratingen
  - Praxis Dr.med. Werner A. Biewer, Saarbrücken
  - Rheumatologische Schwerpunktpraxis am Feuersee, Stuttgart
  - Praxis für Rheumatologie, Ulm